CLINICAL TRIAL: NCT04320238
Title: An Clinic Trial of Recombinant Human Interferon Alpha Nasal Drops to Prevent Coronavirus Disease 2019 in Medical Staff in Epidemic Area
Brief Title: Experimental Trial of rhIFNα Nasal Drops to Prevent 2019-nCOV in Medical Staff
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhongji Meng, Chief of Infectious disease department, Principal Investigator, Clinical Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interferon_prophylaxis
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: 2019 Novel Coronavirus Infection
Keywords: rhINF-α; 2019-nCOV; prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-risk group (Experimental): medical staff work in non-isolated general wards or laboratories, not directly contact with COVID-19 patients.
  Interventions: Drug: recombinant human interferon Alpha-1b
- high-risk group (Experimental): doctors and nurses work in isolated ward, directly contact with COVID-19 patients.
  Interventions: Drug: recombinant human interferon Alpha-1b; Drug: thymosin alpha 1

INTERVENTIONS:
Drug: recombinant human interferon Alpha-1b — recombinant human interferon Alpha-1b nasal drops, 2-3 drops for each nostril per time, 4 times per day.
  Other Names: interferon α
Drug: thymosin alpha 1 — thymosin alpha 1 subcutaneous injection 1 time per week.
  Other Names: thymosin α
  Arms: high-risk group

SUMMARY:
The investigators plan to carry out an experimental study on the preventive effect of recombinant human interferon alpha nasal drops on the infection of 2019 new coronavirus in medical staff.

DETAILED DESCRIPTION:
The investigators plan to carry out an experimental study enrolling more than 2000 medical staff and divide participants into low-risk group and high-risk group according to whether they can directly exposed to 2019-nCOV infected patients. In the low-risk group, participants will be given recombinant human interferon alpha-1b nasal drops (2-3 drops/nostril/ time, 4 times/ day), and in the high-risk group will be given preventive intervention with interferon nasal drops and thymosin-α (thymosin was injected subcutaneously once / week), and the intervention time is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Formally serving medical staff in Taihe Hospital;

Exclusion Criteria:

* pregnant women;
* severe chronic diseases who are unable to participate in daily routine work;
* fever (temperature≥37.3 ° ) and / or respiratory symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2944 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
new-onset COVID-19 | From date of randomization until the diagnosis of COVID-19, assessed up to 6 weeks.
  new-onset coronavirus disease-2019

SECONDARY OUTCOMES:
Number of Participants with coronavirus related symptoms | during 28-day intervention.
  new-onset fever or respiratory symptoms but with negative pulmonary images evidence.
Number of Participants with adverse effect | during 28-day intervention.
  adverse effect of interferon α

CONTACTS AND LOCATIONS:
Locations (1):
- Taihe Hospital, Shiyan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Tang X, Wu C, Li X, Song Y, Yao X, Wu X, Duan Y, Zhang H, Wang Y, Qian Z, Cui J, Lu J. On the origin and continuing evolution of SARS-CoV-2. Natl Sci Rev. 2020 Jun;7(6):1012-1023. doi: 10.1093/nsr/nwaa036. Epub 2020 Mar 3. PMID 34676127
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Thompson R. Pandemic potential of 2019-nCoV. Lancet Infect Dis. 2020 Mar;20(3):280. doi: 10.1016/S1473-3099(20)30068-2. Epub 2020 Feb 7. No abstract available. PMID 32043978